CLINICAL TRIAL: NCT00212849
Title: Autologous Chondrocyte Implantation in the Patellofemoral Joint
Status: Completed | Type: Observational
Sponsor: Orthopaedic Research Foundation (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Other Study IDs: JF_ACIPF091305
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2004-12

CONDITIONS: Chondrosis; Patellar Articular Cartilage Lesions; Trochlear Articular Cartilage Lesions
Keywords: Articular Cartilage Lesions; Patellar lesions; Trochlear lesions; Patellofemoral joint; Carticel; Autologous Chondrocyte Implantation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to measure the outcomes of patients who have articular cartilage lesions in the patellofemoral joint and are treated with the Autologous Chondrocyte Implantation.

DETAILED DESCRIPTION:
Cartilage restoration, in general, is a relatively new option for the treatment of articular cartilage lesions primarily of the knee. In the initial autologous cultured chondrocyte transplantation (ACT or, by others implantation, thus ACI) reported by Peterson et. al., the results of femoral lesions were favorable, while 5 of 7 patellofemoral treatments were poor. In the United States, the expedited FDA approval based on these results excluded the patella. As a result, in the United States, it has been difficult to further evaluate use of ACI at the patellofemoral joint in light of the exclusion of "off label" uses by many governmental and private insurance programs. Nevertheless, a growing body of knowledge is accumulating outside the United States that the use of ACI at the patella is a viable option and soon similar findings will be published in the US by Minas et. al. (accepted for publication)

ELIGIBILITY:
Inclusion Criteria:

* Carticel Implantation of the patella and/or trochlear lesion. Patients who have reached their two-year follow-up date. All patients included in sequential order.

Exclusion Criteria:

* Patients that have had a microfracture in the knee joint at the same time as Carticel Implantation.

Patients that have implantable lesions other than the patella and trochlea.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35
Dates: Start 1995-01; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Jack Farr, MD, Principal Investigator — Orthopaedic Research Foundation, Inc.
Locations (1):
- Orthopaedics Indianapolis, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Minas T, Bryant T. The role of autologous chondrocyte implantation in the patellofemoral joint. Clin Orthop Relat Res. 2005 Jul;(436):30-9. doi: 10.1097/01.blo.0000171916.40245.5d. PMID 15995417